CLINICAL TRIAL: NCT02971852
Title: Hypnotic Glove Anesthesia: Effects of Hypnosis on Skin Temperature Measured by Infrared Thermography
Brief Title: Effects of Hypnosis on Skin Temperature
Status: Completed | Type: Observational
Sponsor: Claude Bernard University (Other)
Collaborators: Centre Clinical, France (Other); Saint-Gregoire Private Hospital Center (Other); Institut Émergences, France (Unknown)
Responsible Party: Principal Investigator, Emmanuel Boselli, MD, PhD, Claude Bernard University
Other Study IDs: Hypnotic glove anesthesia
Record Dates: First submitted 2016-11-15; First posted 2016-11-23 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Hypnosis; Healthy Volunteers
Keywords: Hypnosis; Anesthesia; Suggestion; Thermography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypnotic glove anesthesia is a hypnosis technique wherein the patient, following the suggestions of the hypnotherapist, is mentally capable to create a loss of sensation in areas of the hand that would be covered by a glove. We investigated the effects of hypnotic glove anesthesia on skin temperature measured by thermography.

DETAILED DESCRIPTION:
After 20 min installation and temperature equilibration (T0), the subject skin temperature was recorded in 5 regions of both hands (1 = distal hand, 2 = proximal hand, 3 = wrist, 4 = distal forearm, 5 = proximal forearm) using infrared thermography.

After 10 min of latency, skin temperature was recorded again in both hands (T1).

A first noxious stimulus (NOX1) is then applied by the hypnotherapist by pinching the webbing between the thumb and index fingers of the dominant hand between the thumb and the index. Pain intensity is assessed on a 0-10 (0 = no pain, 10 = maximal pain imaginable) numerical rating scale (NRS1).

The hypnotic glove is then mentally created by the subject on his dominant hand following the suggestions of the hypnotherapist (T2). To assess the efficacy of the hypnotic glove, a second noxious stimulus (NOX2) is applied similarly to NOX1 and the NRS was recorded (NRS2).

The subject is then invited to mentally wear off the glove (T3). Skin temperature is then recorded in both hands, and a third noxious stimulus (NOX3) is applied similarly to NOX1 and NOX2 to verify the disappearance of hypnotic anesthesia.

A last record of skin temperature in both hands is performed 5 min after the glove is withdrawn (T4).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged from 18 to 75

Exclusion Criteria:

* Neurologic or psychiatric disorder
* Upper limb amputation
* Microcirculation abnormalities (e.g. Raynaud syndrome)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in skin temperature during the experiment in the hand and forearm | During the study experiment, from the beginning of the experiment, after 20 min installation and temperature equilibration, to the end of the experiment, 5 min after the glove is mentally withdrawn (approximately 1 h).
  Comparison of skin temperature between the dominant ("wearing" the hypnotic glove) and the non-dominant hand and forearm in the 5 predefined regions from Time 0 to Time 4.

SECONDARY OUTCOMES:
Change in pain intensity during the experiment following noxious stimulation | During the study experiment, from 10 min after the beginning of the experiment to 5 min before the end of the experiment, when the glove is mentally withdrawn (approximately 45 min).
  Comparison of pain intensity following noxious stimulation assessed by 0-10 NRS scale at Time 1, Time 2 and Time 3 in the dominant hand ("wearing" the hypnotic glove).

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Paqueron, MD, PhD, Principal Investigator — Centre Clinical, France
Locations (3):
- France (3):
  - Institut Émergences, Rennes
  - Centre hospitalier privé Saint-Grégoire, Saint-Grégoire
  - Centre Clinical, Soyaux

IPD SHARING:
Plan to Share IPD: No